CLINICAL TRIAL: NCT02736396
Title: Southend Imaging Study
Acronym: SIS
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: P0867
Record Dates: First submitted 2016-03-08; First posted 2016-04-13 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Cognition Disorders
MeSH Terms: conditions — Cognition Disorders | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Medical History, Neuropsychological tests, clinical assessments, fMRI
  Interventions: Other: fMRI; Other: Neuropsychological tests
- Cognitive impairment: Medical History, Neuropsychological tests, clinical assessments, fMRI
  Interventions: Other: fMRI; Other: Neuropsychological tests

INTERVENTIONS:
Other: fMRI — Functional MRI scan to be performed
Other: Neuropsychological tests — Cognitive assessments will be performed, including Mini Mental State Examination, Rey Auditory Verbal Learning Test, Stroop, Visual Short Term Memory Assessment.

SUMMARY:
The study objective is to correlate global cognition and episodic memory performance to resting state fMRI functional connectivity. This is a non-treatment, prospective, natural history data collection study in a cross-sectional cohort of patients with cognitive impairment.

DETAILED DESCRIPTION:
At present, Magnetic Resonance Imaging (MRI) is widely used along with other tests to help diagnose dementia, however diagnosis still remains challenging. There is currently a focus on the usefulness of resting state functionalMRI (RS fMRI) as a way of establishing differences in functional connectivity between healthy subjects and those with various neurodegenerative disorders. Although the potential for RS fMRI to be used as a biomarker for neurological diseases looks promising, further research is needed, especially regarding validation of normal values and seed-based functional connectivity. Further research into this area will help to improve the ability to appropriately classify new subjects and ultimately allow use of RS functional connectivity as a biomarker. This is a nontreatment, prospective, natural history data collection that aims to analyse functional connectivity in a cohort of patients with suspected cognitive impairment. Correlation of global cognition and episodic memory performance to resting state fMRI functional connectivity will be evaluated. Patient population will include patients over the age of 18 with cognitive impairment and age and gender matched controls. Eligible patients will have to complete neuropsychological and clinical assessments and complete an fMRI scan prior to enrolment.Study duration is estimated at 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Cognitive impairment
* Age from 18 to 100 years
* On stable medication for 1 month before the screening visit; on or off cholinesterase inhibitors
* Fluency in English and adequate premorbid intellectual functioning

Exclusion Criteria:

* Any contraindication to MRI scanning
* Clinically significant psychiatric disorder (e.g. depression)
* Current clinically significant illness that could confound the results of the study
* History of alcohol or drug dependence or abuse
* Current use of anticonvulsant or narcotic medications.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with suspected cognitive impairment, mild cognitive impairment, autosomal dominant Alzheimer's disease, late onset Alzheimer's disease, Vascular dementia, Parkinson's dementia and age and gender matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the functional connectivity in the Default Mode Network . | 4 years
  Evaluating the correlation of the Default Mode Network functional connectivity to types of dementia.

SECONDARY OUTCOMES:
Correlation of cognitive performance to functional connectivity. | 4 years
  To evaluate the correlation between individual measures of functional connectivity and global and episodic cognitive performance as measured by neuropsychological tests.

CONTACTS AND LOCATIONS:
Overall Officials: Paula A Harman, BSc, Principal Investigator — Southend University Hospital NHS Foundation Trust
Locations (1):
- Southend Hospital, Westcliff-on-Sea, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No